CLINICAL TRIAL: NCT07186231
Title: Comparative Effects of Blood Flow Restriction and Traditional Strength Training on Proximal Shoulder Musculature: A Randomized Clinical Trial
Brief Title: Strength Training With and Without Blood Flow Restriction on Shoulder Muscle Strength in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alice Maria da Costa Carvalhais (Other)
Responsible Party: Sponsor-Investigator, Alice Maria da Costa Carvalhais, Auxiliary Professor, Cooperativa de Ensino Superior, Politécnico e Universitário
Organization: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31/CE-IPSN/2024
Record Dates: First submitted 2025-09-07; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Resistance Training; Blood Flow Restriction (BFR) Training Effects
Keywords: Resistance training; Blood Flow Restriction; Hypertrophy; Strength; Power; Endurance
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-load strength training with Blood Flow Restriction (Experimental): Participants allocated to this study arm, performed a 4-week training with 2 sessions per week, using low load resistance training with Blood Flow Restriction.
  Interventions: Device: Low-load resistance training with Blood flow Restriction
- High-load strength training (Active Comparator): Participants allocated to this study arm performed 4-week training with 2 sessions per week, using high-load resistance training.
  Interventions: Other: High-load resistance training.

INTERVENTIONS:
Device: Low-load resistance training with Blood flow Restriction — Each session began with a warm-up including mobility and stretching exercises for the shoulders and upper limbs. During the first session, the one-repetition maximum (1RM) for each participant and exercise was determined using a failure-to-repetition method with applied coefficients. Training was performed at 30 percent 1RM, following a standardized sequence of three shoulder-targeted exercises (shoulder abduction, external rotation, Dumbbell Overhead Press), totaling 75 repetition per session (30/15/15/15), 30-second rest intervals per sets. Movements were executed at a controlled 4-sec. tempo (2 seconds concentric, 2 seconds eccentric). BFR was applied using pneumatic cuffs, maintained during each exercise, released for 60 seconds between exercises, and reapplied for the next. Participants rated exercise difficulty, including pain, tension, and numbness, using a 0-10 numeric scale, with protocol adjustments or session cancellation if symptoms exceeded 7/10.
  Arms: Low-load strength training with Blood Flow Restriction
Other: High-load resistance training. — Each session began with a warm-up including mobility and stretching exercises for the shoulders and upper limbs. During the first session, the 1RM for each participant and exercise was determined using a failure-to-repetition method with applied coefficients. Training was performed at 70 percent following a standardized sequence of three shoulder-targeted exercises (shoulder abduction and external rotation, and Dumbbell Overhead Press). Four sets of 8 to 10 repetitions were completed for each exercise, with 2-minutes rest between sets and exercises. Movement speed was moderate (1-second concentric, 2-second eccentric).
  Arms: High-load strength training

SUMMARY:
The goal of this clinical trial is to compare two types of shoulder strength training: low-load training with blood-flow restriction (BFR) and high-load training without BFR. The study includes healthy adults.

The main questions it aims to answer are:

Are changes in shoulder strength, power, endurance, and muscle mass similar with low-load BFR and high-load training?

Researchers will compare strength training with BFR to strength training without BFR to see whether changes in shoulder muscle performance are similar.

Participants will:

* Provide basic personal details, body measurements (e.g., height and weight), and a brief medical history before starting.
* Train in one of the two programs (BFR or no BFR) two times per week for 4 weeks.
* Complete tests of shoulder maximum strength, power, endurance, and muscle mass at the start and at the end of the protocol.

DETAILED DESCRIPTION:
All outcome assessments were conducted after a standardized warm-up to minimize measurement variability. The warm-up comprised light aerobic activity, followed by dynamic mobility exercises for the shoulder girdle and upper limbs, and targeted stretching of the shoulder and elbow/forearm muscle groups (two sets of 20-30 seconds per muscle group). Safety procedures included monitoring for adverse symptoms during testing and training; sessions were paused or discontinued according to predefined criteria.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18.5 and 30 kg/m²

Exclusion Criteria:

* participation in sports that heavily involve the dominant arm (e.g., tennis, volleyball, or handball) and do not engage in strength training exercises on the upper limb;
* history of trauma or surgery affecting the dominant upper limb;
* acute or chronic shoulder pain,;
* radiating pain;
* cervical disc herniation;
* previous neck surgeries,;
* upper limb edema;
* history of deep vein thrombosis;
* history of oncologic or metabolic conditions;
* pregnancy;
* experience of persistent symptoms such as numbness, tingling, or pain exceeding 7/10 on a numeric scale during the training (applicable to BFR group);
* missed more than one session during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Deltoid muscle mass | Baseline and between 24 hours and 1 week after completion of the 4-week intervention.
  Arm circumference at the armpit level of the dominant limb, used as a proxy for deltoid muscle mass.
Change in shoulder muscle power | Baseline and between 24 hours and 1 week after completion of the 4-week intervention.
  Shoulder muscle power, assessed by the Single Arm Seated Shot-Put Test
Change in shoulder muscle maximal strength | Baseline and between 24 hours and 1 week after completion of the 4-week intervention.
  Maximal isometric muscle strength measured with the Smart Groin Trainer dynamometer (NeuroExcellence, Braga, Portugal) during a vertical lift task.
Change in muscle shoulder endurance | Baseline and between 24 hours and 1 week after completion of the 4-week intervention.
  Shoulder muscle endurance, assessed by the Shoulder Endurance Test (SET)

SECONDARY OUTCOMES:
Change in Numeric Rating Scale | Continuously from the start to the end of each training session, across all sessions during the 4-week intervention (participants report immediately if symptoms reaches ≥7/10.
  Participants in the Low-load strength training with BFR group rate pain, numbness and tingling in the dominant upper limb on a 0-10 Numeric Rating Scale (NRS) (0 = none; 10 = worst imaginable). Sessions are paused if NRS ≥ 7/10.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Carvalhais, PhD, Principal Investigator — Cooperativa de Ensino Superior, Politécnico e Universitário
Locations (1):
- Escola Superior de Tecnologias da Saúde do Tâmega e Sousa, Gandra, Paredes, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT07186231/Prot_SAP_000.pdf